CLINICAL TRIAL: NCT00416975
Title: Breast Cancer Risk-Tailored Messages for More Women
Brief Title: Individualized Risk-Based Education in Promoting Breast Cancer Screening in Healthy Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: MCC-00036; P30CA016059 (NIH); MCC-00036 (Other: Massey Cancer Center)
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Counseling; Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Breast Cancer Risk Assessment Screening (Other): Counseling Intervention and Eduation Intervention
  Interventions: Other: counseling intervention; Other: educational intervention; Procedure: evaluation of cancer risk factors

INTERVENTIONS:
Other: counseling intervention — Women in the intervention group will be offered breast cancer risk assessment at baseline. Computerized risk assessment is followed by personalized risk tailored health messages. The health messages will also include appropriate recommendations for genetic and psychosocial counseling. Baseline measurements from a questionnaire given prior to the intervention will capture current breast cancer screening practices (mammography, clinical breast exam and self exam), intentions to get mammograms, family discussion of breast cancer, risk perceptions, and breast cancer worry. Important demographic variables and breast cancer risk factors will also be measured. Participants will receive follow up telephone interviews at 1, 6, and 18 months to assess mammography use.
Other: educational intervention — Women in the intervention group will be offered breast cancer risk assessment at baseline. Computerized risk assessment is followed by personalized risk tailored health messages. The health messages will also include appropriate recommendations for genetic and psychosocial counseling. Baseline measurements from a questionnaire given prior to the intervention will capture current breast cancer screening practices (mammography, clinical breast exam and self exam), intentions to get mammograms, family discussion of breast cancer, risk perceptions, and breast cancer worry. Important demographic variables and breast cancer risk factors will also be measured. Participants will receive follow up telephone interviews at 1, 6, and 18 months to assess mammography use.
Procedure: evaluation of cancer risk factors — Women in the intervention group will be offered breast cancer risk assessment at baseline. Computerized risk assessment is followed by personalized risk tailored health messages. The health messages will also include appropriate recommendations for genetic and psychosocial counseling. Baseline measurements from a questionnaire given prior to the intervention will capture current breast cancer screening practices (mammography, clinical breast exam and self exam), intentions to get mammograms, family discussion of breast cancer, risk perceptions, and breast cancer worry. Important demographic variables and breast cancer risk factors will also be measured. Participants will receive follow up telephone interviews at 1, 6, and 18 months to assess mammography use.

SUMMARY:
RATIONALE: Education, based on a patient's risk factors, may help promote breast cancer screening in healthy women.

PURPOSE: This randomized clinical trial is studying individualized risk-based education to see how well it promotes breast cancer screening in healthy women compared to standard education.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the impact of risk-tailored messages vs standard health information on the outcome of mammography in healthy women.

Secondary

* Compare the effect of these interventions on breast self-examination, clinical breast exam, risk perceptions, and breast cancer worry.
* Compare the mechanism of action of these interventions on participants by assessing the impact of covariants (coping mechanisms, expanded Health Belief Model variables, breast cancer worry, breast cancer risk factors including family history, risk perceptions, discussion of breast cancer with relatives, previous screening practices, intentions to screen, and various demographic variables-age, race, and education) on breast cancer screening.

OUTLINE: This is a randomized study.

Participants are approached to complete a baseline survey while they are waiting for their clinic visits. Baseline surveys measure breast cancer risk factors, current breast cancer screening practices, intentions to screen, risk perceptions, breast cancer worry, coping mechanisms, and discussion of breast cancer with relatives. After completion of the baseline surveys, participants are then randomized to 1 of 2 education arms.

* Arm I (intervention group): Participants undergo a computerized risk assessment followed by personalized risk-tailored health messages. Health messages are based on principles of the expanded Health Belief Model (HBM). These messages include screening and lifestyle recommendations, information on the seriousness of breast cancer, instructions on how to arrange a mammography appointment, and contact information for genetic and psychosocial counseling.
* Arm II (control group): Participants receive generalized breast health information sheets that contain appropriate screening and lifestyle recommendations for the general public and contact information for genetic and psychosocial counseling.

All participants undergo follow-up assessment by telephone (or by mail if unreachable by phone) at 1, 6, and 18 months after the initial intervention. Self-reported mammography use, additional breast health monitoring practices, risk perception, breast cancer worry, coping mechanisms, HBM-related beliefs, and family communication are measured.

PROJECTED ACCRUAL: A total of 900 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Receiving care at the Women's Health Center gynecology clinic in downtown Richmond, VA or at either the satellite Stony Point or Hayes Willis clinics
* No history of breast cancer, including in situ lesions
* At least 7 years old at first menarche
* No prior genetic counseling or genetic testing for breast cancer
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* Not pregnant

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 899 (Actual)
Dates: Start 2000-05; Primary Completion 2005-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To reduce the impact of breast cancer by promoting screening, increasing breast health awareness, and providing supportive resources to women who want them; | 12 years

CONTACTS AND LOCATIONS:
Overall Officials: Joann N. Bodurtha, MD, MPH, Principal Investigator — Massey Cancer Center